CLINICAL TRIAL: NCT06313996
Title: A Global Randomized Multicenter Phase 3 Trial to Compare the Efficacy and Safety of Lisocabtagene Maraleucel (JCAR017/BMS-986387) to Standard of Care in Adults With Relapsed or Refractory Follicular Lymphoma (TRANSFORM FL)
Brief Title: A Study to Evaluate the Efficacy and Safety of Liso-cel Compared to Standard of Care in Adults With Relapsed or Refractory Follicular Lymphoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Juno Therapeutics, Inc., a Bristol-Myers Squibb Company (Industry)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CA082-011; 2023-507477-18 (EudraCT Number)
Record Dates: First submitted 2024-02-26; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Relapsed or Refractory Follicular Lymphoma
Keywords: Lisocabtagene Maraleucel; Liso-cel; Follicular Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, Follicular | interventions — Cyclophosphamide; Doxorubicin; Vincristine; Rituximab; Prednisone; Bendamustine Hydrochloride; Lenalidomide; fludarabine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): Active Comparators:
  R-CHOP (rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone)
  B-R (bendamustine and rituximab)
  R2 (rituximab and lenalidomide)
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Rituximab; Drug: Prednisone; Drug: Bendamustine; Drug: Lenalidomide
- Arm B (Experimental): Lisocabtagene Maraleucel
  Interventions: Drug: Fludarabine; Drug: Liso-cel

INTERVENTIONS:
Drug: Cyclophosphamide — Specified dose on specified days
  Arms: Arm A
Drug: Doxorubicin — Specified dose on specified days
  Arms: Arm A
Drug: Vincristine — Specified dose on specified days
  Arms: Arm A
Drug: Rituximab — Specified dose on specified days
  Arms: Arm A
Drug: Prednisone — Specified dose on specified days
  Arms: Arm A
Drug: Bendamustine — Specified dose on specified days
  Arms: Arm A
Drug: Lenalidomide — Specified dose on specified days
  Arms: Arm A
Drug: Fludarabine — Specified dose on specified days
  Arms: Arm B
Drug: Liso-cel — Specified dose on specified days
  Other Names: Lisocabtagene Maraleucel; BREYANZI
  Arms: Arm B

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Liso-cel compared to standard of care in adults with Relapsed or Refractory Follicular Lymphoma.

DETAILED DESCRIPTION:
The purpose of this phase III study is to evaluate the clinical benefit of liso-cel for the treatment of r/r FL by comparing it to standard of care therapy in patients with r/r FL, with progression-free survival (PFS) as the primary endpoint.

The primary objective is to demonstrate superiority of the Liso-cel treatment strategy over standard of care (SOC) therapy with respect to progression-free survival (PFS) determined by independent review committee (IRC) based on the Lugano response criteria.

Participants randomized to Arm A (Standard of Care) will receive RCHOP, BR, or R2 based on investigator choice and this has to be determined prior to randomization.

Participants randomized to Arm B (Liso-cel treatment) will receive a single infusion CAR-positive viable T-cells.

ELIGIBILITY:
Inclusion Criteria

* Participants must have measurable disease.
* Participants must have previously been treated with certain defined anti-cancer therapies and their disease must have come back or must have not responded to the previous or last treatment.
* Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Participants that have histologically confirmed Follicular Lymphoma (FL) (Grade 1, 2, or 3a) corresponding to the most recent relapse prior to screening.
* Participants that have Relapsed or refractory FL, as assessed by the Investigator.
* Participants that have received at least one prior line and no more than three prior lines of systemic therapy including a combination of an anti-CD20 antibody and an alkylating agent.
* Participants that received one prior line of systemic therapy are eligible if they present with high risk features.

Exclusion Criteria

* Participants must not have any history of heart problems.
* Participants must not have any bleeding disorders.
* Participants must not have any Central Nervous System involvement by Follicular Lymphoma or other brain conditions.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-03-29 (Estimated); Primary Completion 2031-10-16 (Estimated); Study Completion 2031-10-16 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Up to 5 years from the last participant randomized
  Defined as the time from randomization to death due to any cause or progressive disease (PD) per independent review committee (IRC) assessment using the Lugano 2014 Criteria, whichever occurs first

SECONDARY OUTCOMES:
Complete response (CR) | Up to 5 years from the last participant randomized
  Defined as participants achieving a complete response per IRC assessment using the Lugano 2014 Criteria
Overall survival (OS) | Up to approximately 7 years
  Defined as the time from randomization to death due to any cause
Overall response (OR) | Up to 5 years from the last participant randomized
  Defined as participants achieving a response (CR or partial response (PR)) per IRC assessment using the Lugano 2014 Criteria
Duration of response (DOR) | Up to 5 years from the last participant randomized
  Defined as the time from first response (CR or PR) per IRC assessment using the Lugano 2014 Criteria to PD or death due to any cause, whichever occurs first
Event-free survival (EFS) | Up to 5 years from the last participant randomized
  Defined as the time from randomization to the first documentation of progressive disease (PD) per IRC assessed using the Lugano 2014 Criteria start of new anti-cancer therapy, or death due to any cause, whichever occurs first
Time to next anti-cancer therapy (TTNLT) | Up to 5 years from the last participant randomized
  Defined as time from randomization to start of new anti-cancer therapy or death due to any cause, whichever occurs first
PFS rate | Up to 5 years from the last participant randomized
EFS rate | Up to 5 years from the last participant randomized
OS rate | Up to approximately 7 years
Progression-free survival on the next line of treatment (PFS-2) | Up to 5 years from the last participant randomized
  Defined as the time from randomization to death from any cause or tumor progression on next line treatment per Investigator assessment, whichever occurs first
Number of participants with adverse events (AEs) | Up to 5 years from the last participant randomized
Number of participants with adverse event of special interest (AESIs) | Up to 5 years from the last participant randomized
Number of participants with serious adverse events (SAEs) | Up to 5 years from the last participant randomized
Number of participants with laboratory abnormalities | Up to 5 years from the last participant randomized
Frequency and length of hospitalizations | Up to 5 years from the last participant randomized
Number of participants with intensive care unit (ICU) inpatient days | Up to 5 years from the last participant randomized
Number of participants with non-ICU inpatient days | Up to 5 years from the last participant randomized
Mean change from baseline in key health-related quality of life (HRQoL) domains. | Up to 5 years from the last participant randomized
  Key HRQoL Domains:
  Global health status/quality of life (GHS/QoL), fatigue, pain, physical functioning, role functioning, cognitive functioning from The European Organization for Research and Treatment of Cancer - Quality of Life C30 Questionnaire (EORTC QLQ C30), and Symptom Burden and Physical Condition/Fatigue from the European Quality of Life Module Non-Hodgkin's Lymphoma Low-Grade 20 items (EORTC QLQ-NHL-LG20)
Time to meaningful improvement/deterioration in key HRQoL domains. | Up to 5 years from the last participant randomized
  Key HRQoL Domains:
  Global health status/quality of life (GHS/QoL), fatigue, pain, physical functioning, role functioning, cognitive functioning from The European Organization for Research and Treatment of Cancer - Quality of Life C30 Questionnaire (EORTC QLQ C30), and Symptom Burden and Physical Condition/Fatigue from the European Quality of Life Module Non-Hodgkin's Lymphoma Low-Grade 20 items (EORTC QLQ-NHL-LG20)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm